CLINICAL TRIAL: NCT05168319
Title: Effects and Mechanism of Prolonged Continuous Theta Burst Stimulation on Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-0751
Record Dates: First submitted 2021-12-15; First posted 2021-12-23 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2022-01

CONDITIONS: Neuropathic Pain; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Neuralgia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: fifty NP patients were randomly assigned to 3 groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and assessors were blind to group assignment until the study was completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pcTBS (Experimental): pcTBS was administered to the left M1 at 80% resting motor threshold (RMT), consisting of a burst of 3 pulses given at 50 Hz repeated every 5 Hz. A total of 1,200 pulses were delivered with the TMS coil positioned in a posterior-anterior (PA) direction parallel to the midline.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- 10HZ rTMS (Active Comparator): The rTMS protocol included 15 trains of 10-second stimulation given at 10 Hz to the left M1 at 80% resting motor threshold (RMT), with the inter-train interval being set to 50 seconds (1500 pulses)
  Interventions: Device: Repetitive transcranial magnetic stimulation
- Sham (Sham Comparator): The Sham stimulation was delivered using the same protocol, with the coil being orientated at 90° to the scalp so that the magnetic field would be delivered away from the scal
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Participants received 10HZ rTMS protocol consisted of 5 sessions over 5 consecutive workdays
  Arms: 10HZ rTMS
Device: Repetitive transcranial magnetic stimulation — Participants received pcTBS protocol consisted of 5 sessions over 5 consecutive workdays
  Arms: pcTBS
Device: Sham stimulation — Participants received Sham rTMS stimulations consisted of 5 sessions over 5 consecutive workdays
  Arms: Sham

SUMMARY:
Neuropathic pain (NP) is one type of refractory chronic pain condition,medical treatments for NP is limited because of its poorly response. A noninvasive brain-stimulation method called transcranial magnetic stimulation (TMS) has garnered interest as an alternative treatment for intractable NP potentially through inducing therapeutic brain plasticity.Indeed, high-frequency (≥ 5 Hz) Repetitive TMS (rTMS) over the primary motor cortex (M1) is suggested to be able to reduce neuropathic pain in randomized controlled studies.Overall, the clinical application of rTMS in chronic pain is still limited by the response rate,the investigation of rTMS protocols is important for improving rTMS analgesia. Theta burst stimulation (TBS) mimics the bursts of neuronal firing which results in robust long-term potentiation. Continuous TBS (cTBS) is designed to decrease excitability, whereby prolonged cTBS (pcTBS, i.e. multiple cTBS being delivered continuously) has recently been demonstrated to increase excitability. More importantly, pcTBS was found to have comparable or even better analgesic effects than standard 10 Hz rTMS. These findings together call for more studies to validate the analgesic efficacy of pcTBS.

In this study, the investigators aim to assess and compare the efficacy of prolonged continuous theta burst stimulation (pcTBS) with 10HZ rTMS in NP patients.

DETAILED DESCRIPTION:
The investigators designed a randomized, double-blind, sham-controlled study at 1 center. fifty NP patients were randomly assigned to 3 groups. A series of 5 daily pcTBS(1200 pulses/session) or 10-Hz rTMS (1500 pulses/session) of primary motor cortex (M1) or sham stimulation was applied to each patients.

ELIGIBILITY:
Inclusion Criteria:

* (1)woman or man over 18 and under 70 years old; （2）pain fulfilling the criteria for probable or definite peripheral neuropathic pain ; (3) pain for at least 3 months, continuous pain (at least four days per week), at least moderate intensity (≥ 4/10 assessed by VAS) ; (4) stable pharmacological treatment for pain at least 2 weeks before inclusion; (5) able to cooperate in completing questionnaire.

Exclusion Criteria:

* (1) Any clinically significant or unstable ongoing medical or psychiatric disorder including major depression; (2) History of substance abuse (alcohol, drugs); (3) Past treatment with repetitive transcranial magnetic stimulation (rTMS); (4) Contraindications to rTMS (previous severe head trauma or neurosurgical intervention, past or current epilepsy, active brain tumor, intracranial hypertension, implanted ferromagnetic devices, e.g., cardiac pacemaker, neurostimulator, or cochlear implants); (5) other type of pain more severe than neuropathic pain; (6) Any difficulty to fill out questionnaires (due to language or cognitive problems); (7) impossibility to be followed during the time course of the study;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
The mean change from baseline in pain intensity measured with the visual-analogic scale (VAS) | through study completion, an average of 8 months
  The primary outcome measure was the mean change from baseline over the course of 5 (group by time interaction) in average pain intensity measured with the visual-analogic scale (VAS) ( 0= no pain and 10= maximal pain). Baseline average pain intensity was assessed at inclusion then on the day of randomization, just before the first rTMS session (day 1) and corresponded to the average of these two values.

SECONDARY OUTCOMES:
Motor-evoked potential (MEP) | through study completion, an average of 8 months
  Corticospinal excitability was measured with MEP at rest of the first dorsal interosseous (FDI) muscle, A total of 20 single pulses were consecutively delivered to the hand region of the left M1 at 120% RMT (45° to the midline, handle pointing backward).
Cortical silent period (CSP) | through study completion, an average of 8 months
  Corticospinal excitability was measured with CSP during a sustained voluntary FDI muscle contraction, A total of 20 single pulses were consecutively delivered to the hand region of the left M1 at 120% RMT (45° to the midline, handle pointing backward).
The sensory dimension of pain and affective dimension of pain | through study completion, an average of 8 months
  The sensory dimension of pain (rated on 33) and affective dimension of pain (rated on 12) from the 15-items Short form of the McGill Pain questionnaire (SF-MPQ) .
Pain interference scale | through study completion, an average of 8 months
  7 items rated from 0= does not interfere to 10= complete interference, total score 70 from the Brief Pain Inventory.
Patients global impression of change | through study completion, an average of 8 months
  the 7 items Patients global impression of change (PGIC) (from very much worse to very much improved)
The depression score | through study completion, an average of 8 months
  ranging from 0 to 13 with higher scores indicating more severe depression from the 13 items Beck Depression Inventory (BDI)
release of neurotransmitters | through study completion, an average of 8 months
  Measured with magnetic resonance spectroscopy,MRS

CONTACTS AND LOCATIONS:
Overall Officials: min yan, prof, Study Chair — The second affiliated hospital of Zhejiang University hangzhou
Locations (1):
- The second affiliated hospital of Zhejiang University hangzhou, Hangzhou, Zhejiang, China